CLINICAL TRIAL: NCT01234649
Title: Effects of Intervention With the Glucagon-like Peptide 1 (GLP-1) Analog Liraglutide Plus Metformin Versus Metformin Monotherapy in Overweight/Obese Women With Metabolic Defects and Recent History of Gestational Diabetes Mellitus (GDM)
Brief Title: Combined Liraglutide and Metformin Therapy in Women With Previous Gestational Diabetes Mellitus (GDM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Woman's (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Karen Elkind-Hirsch, Scientific Director of Research, Woman's
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RP10-012
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Gestational Diabetes Mellitus; Type 2 Diabetes Mellitus; Metabolic Syndrome; Impaired Glucose Tolerance; Disorder of Glucose Regulation
Keywords: gestational diabetes mellitus; type 2 diabetes mellitus; metabolic dysfunction; impaired fasting glucose; impaired glucose tolerance; incretin mimetic
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Metabolic Syndrome; Glucose Intolerance | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin XR plus liraglutide (Experimental): Metformin XR plus Liraglutide Metformin extended release (XR) 500 mg qd 2 weeks 500 mg bid 2 weeks 500 mg am, 1000 mg pm- 2 weeks 1000 mg bid- 84 weeks (end study) Liraglutide - start .6 mg SC QD step up to 1.2 mg to a max dose of 1.8 mg SC QD as tolerated
  Interventions: Drug: Metformin XR plus liraglutide
- Metformin XR plus placebo (Active Comparator): Metformin plus Placebo Metformin 500 mg qd 2 weeks 500 mg bid 2 weeks 500 mg am, 1000 mg pm- 2 weeks 1000 mg bid -84 weeks (end study) Placebo-start 1 injection SC QD step up to a max dose as tolerated
  Interventions: Drug: Metformin XR plus placebo

INTERVENTIONS:
Drug: Metformin XR plus placebo — Metformin plus Placebo Metformin 500 mg qd 2 weeks 500 mg bid 2 weeks 500 mg am, 1000 mg pm- 2 weeks 1000 mg bid -98 weeks (end study) Placebo-start 1 injection SC QD step up to a max dose as tolerated
  Other Names: Metformin XR is generic
  Arms: Metformin XR plus placebo
Drug: Metformin XR plus liraglutide — Metformin XR-500 qd for 2 weeks, 500 mg bid 2 weeks; 500 mg am, 1000 mg pm- 2 weeks - 1000 bid final dose Liraglutide- start 0.6 mg SC QD step up to 1.2 mg to a max dose of 1.8 mg SC QD as tolerated during the 4-wk non-forced dose-escalation period ( maximum allowed dose of 1.8 mg SC QD)
  Other Names: Victoza
  Arms: Metformin XR plus liraglutide

SUMMARY:
A diagnosis of gestational diabetes mellitus (GDM)has significant implications for the future health of the mother. GDM is often the culmination of years of unrecognized and unmodified diabetes risk factors that lead to overt and occult clinical manifestations during pregnancy. Systematic reviews of older studies conclude that 35-60% women with gestational diabetes will develop type 2 diabetes (DM2) at rates much greater than control groups who did not have glucose intolerance during pregnancy. Liraglutide may potentially delay disease progression in GDM considering the beta -(ß-)cell function improvement in DM2 and ß-cell mass shown to increase in animal models. This study will examine if the addition of liraglutide to metformin therapy is more effective than metformin alone in improving insulin sensitivity and normalizing insulin secretion in at-risk overweight/obese women with prior GDM.

DETAILED DESCRIPTION:
Gestational diabetes is often the culmination of years of unrecognized and unmodified diabetes risk factors that lead to overt and occult clinical manifestations during pregnancy. . Despite the high and increasing rate of type 2 diabetes in Louisiana, the medical community does not have reliable estimates of the number of woman living in southern Louisiana who develop diabetes subsequent to GDM. Systematic reviews of older studies conclude that 35-60% women with gestational diabetes will develop type 2 diabetes at rates much greater than control groups who did not have glucose intolerance during pregnancy. The higher rates were in studies of particular ethnic groups in the U.S. Recently, follow-up programs elsewhere also have identified increasing rates of type 2 diabetes by 5-10 years after GDM: 9-43% type 2 diabetes in Europe and 11-21% in Asia. The frequency of type 2 diabetes is influenced by BMI, weight gain after pregnancy, family history of diabetes, fasting and postchallenge glucose levels during and after pregnancy, postpartum insulin resistance and inadequate β-cell secretion, and the need for pharmacological treatment during pregnancy. However, the risk factors are unable to predict all cases of subsequent type 2 diabetes: the biggest risk factor is a GDM pregnancy. Presently, in the literature, there are described new, more efficient methods of diabetes prevention in groups with a high risk of this disorder, which involve both, lifestyle modification and pharmacological therapies. Lifestyle intervention was found to reduce the incidence of type 2 diabetes by 58% and metformin by 31% as compared with placebo. The use of rosiglitazone in subjects with prediabetes resulted in a 60% reduction of the diabetes incidence rate. Studies are needed for optimal postpartum and long-term health of women who have had GDM. Considerable recent evidence suggests that incretin-based therapies may be useful for the treatment of DM2 because continuous administration of glucagon-like peptide 1 (GLP-1) produces substantial improvements in glucose control and ß-cell function in subjects with type 2 diabetes. Infusion of GLP-1 improves first and second-phase insulin secretion suggesting that early GLP-1 therapy may preserve ß-cell function in subjects with IGT or mild DM2. Whereas native GLP-1 has a very short half-life, the GLP-1 analogue liraglutide has a prolonged action (t1/2=13 h) suitable for once-daily injection. Liraglutide may potentially delay disease progression in GDM considering the ß-cell function improvement in DM2 and ß-cell mass shown to increase in animal models. This study will examine if the addition of liraglutide to metformin therapy is more effective than metformin alone in improving metabolic parameters in at-risk overweight/obese women with prior GDM

ELIGIBILITY:
Inclusion Criteria:

* Adult female 18 years to 45 years of age who experienced GDM within 52 weeks of index pregnancy
* Actual BMI >25 kg/ m2
* Written consent for participation in the study
* Patient completed lactation
* Dysglycemia (impaired fasting glucose [IFG}, impaired glucose tolerance [IGT} or IFG/IGT) and/or ß-cell dysfunction postpartum requiring pharmacological intervention (except type 1 or 2 diabetes)

Exclusion Criteria:

Personal or family history of medullary thyroid carcinoma or in patients with Multiple Endocrine Neoplasia syndrome type 2

* History of pancreatitis
* Significant cardiovascular, cerebrovascular, renal, or hepatobiliary diseases in the past (viral hepatitis, toxic hepatic damage, jaundice of unknown etiology)
* Serum liver enzymes (AST and/or ALT levels) exceeding more than twice normal laboratory values
* Uncontrolled hypertension (systolic blood pressure>150 mm Hg and/or diastolic blood pressure >90 mm Hg)
* Fasting serum triglycerides ≥800 mg/dl at screening. Lipid-lowering medications must have been maintained at the same dose for 3 months prior to enrollment
* Hematological profiles considered to be clinically significant
* Cholestasis during the past pregnancy
* Presence of contradictions for GLP-1 receptor agonist or metformin administration such as allergy or hypersensitivity
* Current use of metformin, thiazolidinediones, dipeptidyl peptidase-4 inhibitors or GLP-1 receptor agonist medications.
* Use of drugs known to exacerbate glucose tolerance.
* Use of prescription or over-the-counter weight-loss drugs
* Diabetes postpartum or history of diabetes or prior use of medications to treat diabetes except gestational diabetes
* Creatinine clearance less than 60 ml/min
* History or currently undergoing chemotherapy or radiotherapy for cancer
* Pregnancy planned during the coming two years
* Currently breastfeeding
* Exclusion criteria include any condition, which in the opinion of the investigator would place the subject at increased risk or otherwise make the subject unsuitable for participation in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2011-08-11 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Elkind-Hirsch, Ph.D., Principal Investigator — Woman's Hospital, Louisiana; Renee Harris, M.D., Study Director — Woman's Hospital, Louisiana
Locations (1):
- Woman's Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elkind-Hirsch KE, Shaler D, Harris R. Postpartum treatment with liraglutide in combination with metformin versus metformin monotherapy to improve metabolic status and reduce body weight in overweight/obese women with recent gestational diabetes: A double-blind, randomized, placebo-controlled study. J Diabetes Complications. 2020 Apr;34(4):107548. doi: 10.1016/j.jdiacomp.2020.107548. Epub 2020 Feb 1. PMID 32046931

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 153 met criteria and were randomized
Pre-assignment Details: 166 were consented but 153 met criteria
Period: Overall Study
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Started | 78 | 75
Completed | 35 | 37
Not Completed | 43 | 38
Not completed — Withdrawal by Subject | 32 | 26
Not completed — Pregnancy | 6 | 6
Not completed — intolerant to side effects | 4 | 3
Not completed — Allergic reaction | 1 | 0
Not completed — Lack of Efficacy | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo | Total
Number analyzed (Participants) | 78 | 75 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 75 | 153
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 75 | 153
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 78 | 75 | 153
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 17 | 28
  White | 67 | 58 | 125
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 78 | 75 | 153
BMI greater than/equal to 25 [Count of Participants; unit: Participants] | 78 | 75 | 153

OUTCOME MEASURES:

1. Primary Outcome: Insulin Secretion-Sensitivity Index (IS-SI)
Description: IS-SI in liraglutide-metformin (LIRA-MET) therapy compared to metformin alone (PLacebo-MET)
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
index | 418.4 (387) | 333 (206)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures design; Test type: Superiority; p < 0.04, ANOVA

2. Secondary Outcome: Fasting Blood Glucose (FBG)
Description: Fasting glucose levels in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
mg/dL | 90 (6.4) | 91.7 (8.4)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p < .005, ANOVA

3. Secondary Outcome: Mean Glucose During OGTT (MBG)
Description: MBG derived from average glucose measured during OGTT in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
mg/dL | 121.6 (20.8) | 118.8 (18.9)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p < 0.011, ANOVA

4. Secondary Outcome: Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: HOMA-IR, a measure of insulin resistance derived from fasting values, in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
index | 2.2 (1.4) | 2.45 (1.5)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Nested repeated measures design; Test type: Superiority; p > 0.05, ANOVA

5. Secondary Outcome: Matsuda Insulin Sensitivity Index Derived From OGTT
Description: OGTT- derived insulin sensitivity index in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
index | 5.9 (2.9) | 5.4 (3.2)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p < 0.03, ANOVA

6. Secondary Outcome: Insulinogenic Index (IGI) /HOMA-IR
Description: IGI/HOMA-IR, a measure of early insulin response corrected by fasting insulin resistance, in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
index | 0.8 (1.14) | 0.62 (0.38)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p > 0.05, ANOVA

7. Secondary Outcome: Absolute Body Weight
Description: Body weight in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
kilograms | 94.2 (18.6) | 91.3 (20)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p < 0.048, ANOVA

8. Secondary Outcome: Change in Body Weight From Baseline to End of Study (Expressed as % Compared to Baseline)
Description: Change in body weight from baseline to end o f study in LIRA-MET group compared with PL-MET group. The number was derived from final weight minus baseline and normalized to a percent.
Time Frame: Change from baseline (time 0) to study end (84 weeks)
Measure: Mean (Standard Error); unit: percent change in weight from baseline
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
percent change in weight from baseline | -7.2 (1.3) | -3.1 (1.4)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Test type: Superiority; p < 0.04, ANOVA

9. Secondary Outcome: Body Mass Index (BMI)
Description: BMI, a measure of total body adiposity, in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: weight (kg) /height (m) squared
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
weight (kg) /height (m) squared | 33.8 (5.2) | 32.8 (6)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p < 0.047, ANOVA

10. Secondary Outcome: Waist Circumference (WC)
Description: Waist size (measure of truncal adiposity) with LIRA-MET compared to PL-MET
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
centimeters | 94.3 (15.2) | 95.3 (15.2)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p < 0.023, ANOVA

11. Secondary Outcome: Waist-to-Hip Ratio (WHR)
Description: Waist circumference divided by hip circumference (a measure of central adiposity) in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: ratio of waist/hip circumference
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
ratio of waist/hip circumference | .81 (.04) | .81 (.05)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p > 0.05, ANOVA

12. Secondary Outcome: Waist to Height Ratio (WHtR)
Description: Waist circumference divided by height (measure of body fat distribution) in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: ratio of waist /height
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
ratio of waist /height | .56 (.08) | .57 (.07)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p = 0.042, ANOVA

13. Secondary Outcome: Total Cholesterol (CHOL) Levels
Description: CHOL levels in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
mg/dL | 183.7 (36) | 183.8 (27)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p > 0.05, ANOVA

14. Secondary Outcome: High Density Lipoprotein Cholesterol (HDL-C) Levels
Description: HDL-C levels in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
mg/dL | 51 (12.6) | 48.7 (11.7)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p > 0.05, ANOVA

15. Secondary Outcome: Low Density Lipoprotein Cholesterol (LDL-C) Levels
Description: LDL-Cholesterol levels in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
mg/dL | 110 (32) | 107 (25)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p > 0.05, ANOVA

16. Secondary Outcome: Triglyceride (TRG) Levels
Description: TRG concentrations in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
mg/dL | 120 (64.5) | 125 (76.4)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p < 0.046, ANOVA

17. Secondary Outcome: Triglyceride to High Density Lipoprotein Cholesterol Ratio TRG/HDL-C)
Description: TRG/HDL-Cholesterol levels in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: ratio of TRG (mg/dL)/HDL-C (mg/dl)
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
ratio of TRG (mg/dL)/HDL-C (mg/dl) | 2.56 (1.5) | 2.95 (2.9)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p < 0.049, ANOVA

18. Secondary Outcome: Systolic Blood Pressure
Description: SBP in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
mmHg | 122 (12) | 123 (12)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p > 0.05, ANOVA

19. Secondary Outcome: Diastolic Blood Pressure
Description: DBP in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
mmHg | 77.6 (8.9) | 77 (9.9)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p > 0.05, ANOVA

20. Secondary Outcome: Alanine Aminotransferase (ALT) Levels
Description: Hepatic enzyme, ALT, associated with insulin resistance, in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
U/L | 32.3 (10.7) | 31 (9.9)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p > 0.05, ANOVA

21. Secondary Outcome: Aspartate Aminotransferase (AST)
Description: The hepatic marker, AST, associated with insulin resistance in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
U/L | 27 (8) | 28 (10.5)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p > 0.05, ANOVA

22. Secondary Outcome: Alanine Aminotransferase /Aspartate Aminotransferase (ALT/AST) Ratio
Description: ALT/AST ratio, used to assess liver function in LIRA-MET group compared with PL-MET group
Time Frame: 84 weeks of treatment
Measure: Mean (Standard Deviation); unit: ratio of ALT (U/L)/ AST (U/L)
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
Number analyzed (Participants) | 35 | 37
ratio of ALT (U/L)/ AST (U/L) | 1.2 (0.4) | 1.18 (0.3)
Statistical Analysis 1: Comparison: Metformin XR Plus Liraglutide vs Metformin XR Plus Placebo; Factorial repeated measures ANOVA; Test type: Superiority; p > 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Data collected over 5 years of trial
Arm/Group | Metformin XR Plus Liraglutide | Metformin XR Plus Placebo
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/75
Other Adverse Events (participants affected / at risk) | 30/78 | 14/75
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin XR Plus Liraglutide (N=78) | Metformin XR Plus Placebo (N=75)
Allergic reaction to liraglutide (Immune system disorders) | 1 (1) | 0 (0) — rash developed at injection site
Nausea (Gastrointestinal disorders) | 29 (29) | 2 (2) — expected side effect of medication
Diarrhea (Gastrointestinal disorders) | 14 (14) | 13 (13) — diarrhea and bloating on higher dose of medication

LIMITATIONS AND CAVEATS:
A large percentage of patients did not complete the trial with the greatest loss from first study visit to second visit. A greater loss was seen initially in the metformin only group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT01234649/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT01234649/ICF_001.pdf